CLINICAL TRIAL: NCT03555539
Title: A Phase 1, 2-Part, Open-Label, Single-Dose, Parallel Group Study to Determine the Effect of Hepatic Impairment on the Safety, Tolerability, and Pharmacokinetics of ACH-0144471 in Adult Subjects
Brief Title: Study of Danicopan in Participants With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ACH471-012
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; Danicopan; ALXN2040; ACH-0144471; Pharmacokinetics; Factor D Inhibitor; Safety
MeSH Terms: interventions — danicopan; rhoA GTP-Binding Protein

STUDY DESIGN:
Intervention Model Description: This study was to be conducted sequentially in 2 parts.
  Part 1: Participants with moderate HI (based on Child-Pugh scores) were compared to demographically matched participants with normal hepatic function.
  Following a review of PK and safety data from Part 1, a decision was to be made by the principle investigators and the sponsor whether to conduct Part 2 of this study, which was planned to enroll participants with severe and mild HI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Healthy Match (Experimental): Single 200-milligram (mg) dose of danicopan on Day 1 in healthy participants (matched control group with normal hepatic function).
  Interventions: Drug: Danicopan
- Part 1: Moderate HI (Experimental): Single 200-mg dose of danicopan on Day 1 in participants with moderate HI.
  Interventions: Drug: Danicopan

INTERVENTIONS:
Drug: Danicopan — Oral tablet.
  Other Names: ALXN2040; ACH-0144471 (formerly); ACH-4471; ACH4471; 4471

SUMMARY:
The purpose of this study was to evaluate the safety, tolerability, and pharmacokinetics (PK) of ACH-0144471 (danicopan) in participants with hepatic impairment (HI) as compared to healthy matched participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index range of 18.0 to 40.0 kilograms (kg)/square meter with a minimum body weight of 50 kg at Screening.
* Females must be of non-childbearing potential.
* Males must agree to abstinence or use a highly effective method of contraception.

HI Participants:

* Be sufficiently healthy for study participation.
* Diagnosis of chronic (>6 months) stable hepatic insufficiency.
* A stable medication regimen.
* In good general health at Screening and check-in, allowing for the concurrent illnesses associated with HI.
* Evidence of cirrhosis due to hepatitis C virus (HCV), hepatitis B virus (HBV) infection, cryptogenic, alcohol abuse, or nonalcoholic steatohepatitis.
* No evidence of hepatocellular carcinoma.
* Have HI as assessed by a Child-Pugh classification score at Screening.

Healthy Participants:

* Participants must be demographically matched to a hepatically impaired participant.
* Medically healthy and without a clinically significant medical history.

Key Exclusion Criteria:

* Evidence of any other clinically significant deviation from normal in a clinical laboratory for the match-controlled participants and laboratory findings beyond those that are consistent with the degree of HI from hepatic participants.
* History of any medical or psychiatric condition or disease.
* Any previous procedure that could alter the absorption or excretion of orally administered drugs.
* Body temperature greater than or equal to 38 degrees centigrade on Day -1 or Day 1 prior to dosing; history of febrile illness or other evidence of infection within 14 days prior to dosing.
* History or presence of drug or alcohol abuse within 6 months prior to dosing; current tobacco/nicotine user; positive for alcohol and/or drugs-of-abuse at Screening or check in.
* Participants who have received eculizumab at any dose or interval within the past 75 days.
* Participation in any other investigational study drug trial 30 days before dosing.
* Donation of whole blood from 3 months before dosing or of plasma from 30 days before dosing; receipt of blood products within 6 months before dosing.

HI Participants:

* Any acute or chronic non-hepatic condition that would limit the participant's ability to participate in this study.
* Any other unspecified reason that would make the participant unsuitable for enrollment.
* Any screening laboratory evaluation outside the laboratory reference ranges not related to HI.
* Fluctuating or rapidly deteriorating hepatic function within the screening period and up to 30 days prior to Day 1.
* History of chronic liver disease due to Wilson's disease.
* History of liver or other solid organ transplants.

Healthy Participants:

* Clinical laboratory evaluations outside of the reference range at Screening or check-in.
* Evidence of acute or chronic liver disease.
* Use of any prescription medications/products within 14 days prior to dosing.
* Use of over-the-counter, nonprescription preparations within 7 days prior to dosing.
* Evidence of chronic HBV or chronic HCV infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Area Under The Plasma Concentration Versus Time Curve From Time 0 Extrapolated To Infinity (AUC0-inf) Of Danicopan | Up to 72 hours postdose
Area Under The Plasma Concentration Versus Time Curve From Time 0 To The Last Measurable Concentration (AUC0-t) Of Danicopan | Up to 72 hours postdose
Maximum Observed Plasma Concentration (Cmax) Of Danicopan | Up to 72 hours postdose
Time To Maximum Observed Plasma Concentration (Tmax) Of Danicopan | Up to 72 hours postdose

SECONDARY OUTCOMES:
Participants Experiencing Treatment-emergent Adverse Events | Day 1 (postdose) through follow-up visit (10 [+/- 2] days after last study drug administration)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes